CLINICAL TRIAL: NCT05300230
Title: Pupillometry Techniques Usage to Quantify the Programming Parameters Effect in the Auditory Effort in Zti Opticon Cochlear Implant Adult Users
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-ZTI-2019-01
Record Dates: First submitted 2020-02-11; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Bilateral Sensorineural Hearing Loss; Unilateral Sensorineural Hearing Loss
Keywords: Bilateral Sensorineural Hearing Loss; Unilateral Sensorineural Hearing Loss; Moderate; Severe; Zti Cochlear implant
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Zti Opticon Cochlear Implant: Patients that are users of Neuro Zti and Neuro 2 processor with a minimum of 6 months of habituation after the implementation.
  Interventions: Device: Neuro Zti cochlear implant and Neuro 2 sound processor

INTERVENTIONS:
Device: Neuro Zti cochlear implant and Neuro 2 sound processor — The study will consist in 3 visits:
  * Visit 1: it will be carried out the first contact and learning the measurement procedure.
  * Visit 2: it will be evaluated the speech perception and the measurement of the pupil dilatation in silence and noise conditions.
  * Visit 3: it will be analysed the effect of the change in the cochlear implant programming parameters.

SUMMARY:
The aim of this study is to establish the connection between the cochlear implant programming parameters with the auditory effort associated with the speech perception evaluated by pupillometry techniques in different audiometric conditions.

ELIGIBILITY:
Inclusion Criteria:

* Users willing to participate in the study with signature and date of the Informed Consent.
* Age between 18 and 70 years old.
* At least 6 months experience with the Neuro Zti implant and Neuro 2 processor.
* Unilateral, bilateral and bimodal users.
* Basic understanding of oral and written Spanish.
* Normal or corrected vision.

Exclusion Criteria:

* Speech or language disorder.
* Added comorbidities or cognitive dysfunction.
* Not approval to participate in the study or absence in some of the programmed sessions for the Cochlear Implant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the Virgen Macarena Hospital of Seville that are users of the Neuro Zti and Neuro 2 processor with at least 6 months of habituation after the implementation.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Analyze the correlation between the speech performance in cochlear implant (CI) users, as measured through the percentage of sentence recognition (%) and the auditory effort, measured by peak pupil dilatation (PPD) in mm. | Up to 12 months after the beginning of the study
  The speech perception will be evaluated through validated sentence recognition tests (such as the HINT test) and the result will be the percentage of correct sentences repeated by the CI patient. The listening effort will be measured through pupillometry techniques in scenarios with different audiometric conditions (different SNR). The result will be the peak pupil dilation in mm.

SECONDARY OUTCOMES:
Evaluate the correlation between the auditory effort as measured through pupillometry techniques and the subjective sensation of the CI patient as rated through validated NASA-TLX questionnaire. | Up to 12-24 months after the beginning of the study
  Analyze the correlation between the objetive auditory effort as measured through pupillometry techniques (peak pupil dilatation, PPD in mm) and the subjetive feeling of effort (fatigue, etc.) as rated by the CI patient in NASA-TLX questionnaire.
Evaluate the correlation between the auditory effort as measured through pupillometry techniques and the cognitive performance of the CI user as measured by different cognitive tests (Nback, Progressive Matrices, Stroop). | Up to 12-24 months after the beginning of the study
  Analyze the correlation between the objetive auditory effort as measured through pupillometry techniques (peak pupil dilatation, PPD in mm) and the cognitive performance of the CI patient as measured through cognitive tests (Nback, Progressive Matrices, Stroop)
Analyze the differences between the auditory effort, as measured through pupillometry techniques in two different CI programming conditions. | Up to 12-36 months after the beginning of the study
  Compare the auditory effort made by the CI patients, as measured by pupillometry techniques, i.e., the peak pupil dilatation (PPD in mm) over two different CI programming conditions: the first condition with the noise filter capability of the CI processor in off mode (VoiceTrack OFF) and the second condition with the noise filters in ON mode (VoiceTrack ON)

CONTACTS AND LOCATIONS:
Overall Officials: Serafín Sánchez Gómez, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain